CLINICAL TRIAL: NCT03830125
Title: A Phase 1, 2-Stage, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BBT-877 Following Single and Multiple Ascending Doses in Healthy Adult Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BBT-877 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bridge Biotherapeutics, Inc. (Industry)
Collaborators: KCRN Research, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBT877-IPF-001
Record Dates: First submitted 2019-01-31; First posted 2019-02-05 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Autotaxin
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — ATX inhibitor BBT-877

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Ascending Doses (Experimental)
  Interventions: Drug: BBT-877, Single dose; Drug: Placebo group
- Multiple Ascending Doses (Experimental)
  Interventions: Drug: Placebo group; Drug: BBT-877, Multiple doses

INTERVENTIONS:
Drug: BBT-877, Single dose — Single dose of BBT-877, 5 dose levels, oral capsule
  Arms: Single Ascending Doses
Drug: Placebo group — Placebo matched to BBT-877, oral capsule
Drug: BBT-877, Multiple doses — Multiple doses of BBT-877, 14 days, 8 dose levels, oral capsule
  Arms: Multiple Ascending Doses

SUMMARY:
This clinical trial is the first-in-human study of BBT-877. The purpose of this phase 1 study is to assess the safety and tolerability of single and multiple ascending oral doses of BBT-877 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and/or female (non-childbearing potential only), 19 to 55 years of age, inclusive, at screening.
* Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dose and throughout the study.
* BMI ≥ 18.5 and ≤ 32.0 kg/m2 and weight ≥ 50 kg at screening.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, as deemed by the PI or designee.
* No clinically significant history or presence of ECG findings as judged by the PI or qualified designee at screening and check-in.
* For a female, must be of non-childbearing potential and therefore must have undergone one of the following sterilization procedures, at least 6 months prior to the first dose:

  1. hysteroscopic sterilization;
  2. bilateral tubal ligation or bilateral salpingectomy;
  3. hysterectomy;
  4. bilateral oophorectomy; or be postmenopausal with amenorrhea for at least 1 year prior to the first dose and follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status.
* A non-vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study drug. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to the first dose of study drug. A male who has been vasectomized less than 4 months prior to the first dose must follow the same restrictions as a non-vasectomized male).
* If male, must agree to not donate sperm from the first dose until 90 days after the last dose of study drug.
* Must have the ability to understand and sign a written informed consent form (ICF), which must be obtained prior to initiation of study procedures.

Exclusion Criteria:

* Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
* History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
* History or presence of alcoholism or drug abuse within the past 2 years prior to the first dose or regular alcohol consumption within 6 months prior to the first dose with an average weekly intake of greater than 21 glasses/units per week for males or 14 glasses/units per week for females, with one unit = 150 mL of wine or 360 mL of beer or 45 mL of 45% alcohol.
* History or presence of hypersensitivity or idiosyncratic reaction to the study drug(s) or related compounds.
* History of anemia or history of decreased red blood cells (RBC).
* Estimated creatinine clearance <80 mL/min at screening.
* Liver function tests (serum ALT, AST, alkaline phosphatase) and serum bilirubin (total and direct) > ULN.
* Baseline hemoglobin, hematocrit, RBC < lower limit of normal at screening and Day -1.
* Female subjects who are pregnant or who are lactating.
* Positive urine drug or alcohol results at screening or check-in.
* Positive urine cotinine at screening.
* Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).
* Unable to refrain from or anticipates the use of:

  * Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements beginning approximately 14 days prior to the first dose and throughout the study. Hormone replacement therapy will not be allowed. After first dosing, acetaminophen (up to 2 g per 24 hours) may be administered at the discretion of the PI or designee.
  * Any drugs known to be significant inducers of CYP3A enzymes and/or P-glycoprotein, including St. John's Wort, for 28 days prior to the first dosing and throughout the study. Appropriate sources (e.g., Flockhart Table) will be consulted to confirm lack of PK/PD interaction with study drug.
* Has been on a diet incompatible with the on-study diet, in the opinion of the PI or designee, within the 28 days prior to the first dose and throughout the study.
* Donation of blood or significant blood loss within 56 days prior to the first dose.
* Plasma donation within 7 days prior to the first dose.
* Exposure to more than four new chemical entities within 12 months prior to first dosing day.
* The subject has participated in a clinical trial and has received an investigational product within 30 days, or 5 half-lives of the investigational product (whichever is longer) of the first dose of study drug in the current study.
* Any condition or circumstance, in the opinion of the PI or designee, which may make the subject unlikely to complete the study or comply with study procedures and requirements, or may pose a risk to the subject's safety.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-11-24 (Actual); Study Completion 2019-11-24 (Actual)

PRIMARY OUTCOMES:
The number and severity of treatment emergent adverse events (TEAEs) | 7 days after the last dose
  To assess the safety and tolerability of single and multiple ascending oral doses of BBT-877 in healthy adult subjects.

SECONDARY OUTCOMES:
Peak Plasma Concentration of BBT-877 in plasma | 72 hours after the last dose
  The PK of BBT-877
Area under the plasma concentration versus time curve of BBT-877 in plasma | 72 hours after the last dose
  The PK of BBT-877
Peak Plasma Concentration of BBT-877 in plasma under fed condition. | 72 hours after the last dose
  The food effect on the PK of a single dose of BBT-877
Area under the plasma concentration versus time curve of BBT-877 in plasma under fed condition. | 72 hours after the last dose
  The food effect on the PK of a single dose of BBT-877
Raw and change-from-baseline values of plasma LPAs | 72 hours after the last dose
  To assess the PD of BBT-877 by assessment of plasma LPAs.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Hyun Ryou, M.D., Ph.D., Study Director — Bridge Biotherapeutics, Inc.
Locations (1):
- Celerion, Lincoln, Nebraska, United States